CLINICAL TRIAL: NCT00203554
Title: Percutaneous Vertebroplasty Versus Conservative Treatment of Pain: A Prospective, Randomized Controlled Study of Osteoporotic Fractures in the Spine
Brief Title: Percutaneous Vertebroplasty Versus Conservative Treatment of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Leif Sorensen, Cons. Neuroradiologist, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20020306
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Pain; Osteoporosis; Fracture
Keywords: osteoporosis; vertebra; fracture; pain; percutaneous; vertebroplasty; polymethylmetacrylate
MeSH Terms: conditions — Pain; Osteoporosis; Fractures, Bone | interventions — Polymethyl Methacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Poly methylmetacrylate, PMMA

SUMMARY:
The purpose of this study is to compare the effect of vertebroplasty with that of traditional medical treatment in the treatment of painful vertebral fractures in osteoporotic patients.

DETAILED DESCRIPTION:
In vertebroplasty a bone cement is injected in one or more fractured vertebra. The indication is pain that needs high doses of analgesics.

The cement is a well known product called poly methyl metacrylate (PMMA) normally used fixate joint prosthesis.

Vertebroplasty is done in local anaesthesia. The treatment was introduced in 1984 in France and today thousands of patients have been treated worldwide, but so far no randomized controlled trials have been published.

ELIGIBILITY:
Inclusion Criteria:

* new pain in spine (within 6 months)
* x-ray verified low energy spinal fracture(s)

Exclusion Criteria:

* less than 20% or more than 90% reduction of the vertebral height
* lack of pain at fracture level
* no need for continuous analgesic treatment
* patient no able to communicate
* general anaesthesia contraindicated
* MRI not possible
* coagulopathy (not adjustable)
* spondylitis
* discitis
* spinal metastasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Level of pain | before treatment and day 1, day 3, day 10 and after 1, 3, 6 and 12 months.

SECONDARY OUTCOMES:
Needs for analgetics, number of days at hospital, level of ADL | before treatment and day 1, day 3, day 10 and after 1, 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Leif Sorensen, Consultant, Principal Investigator
Locations (1):
- Dep of Neuroradiology, Aarhus University Hospital, Aarhus, Denmark